CLINICAL TRIAL: NCT02855281
Title: Sensitivity of PDL-1-analysis From Pleural Effusion in Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: WI_16-233
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC with pleural effusion: The population for selection of potential study participants is comprised of clinical routine patients presenting with (suspected malignant) pleural effusion. These patients must have an indication for pleural puncture. The cause and nature of the pleural effusion at this time point will be unknown in many cases. To establish this, further diagnostic procedures are required. Only patients with confirmed diagnosis of non-small cell lung cancer will be included in the data analysis.

SUMMARY:
This is a prospective diagnostic pilot study to create hypotheses regarding immunocytochemistry (ICC) PD-L1 analysis of pleural effusions in NSCLC patients as compared to the reference standard of PD-L1 immunohistochemistry (IHC). This comparison will be done to assess sensitivity and specificity of PD-L1 detection by ICC in pleural effusions.

ELIGIBILITY:
Inclusion Criteria:

* Presence of malignant pleural effusion with indication for pleural puncture and thoracoscopy
* Confirmed diagnosis of non-small cell lung cancer according to ERS guidelines
* Written informed consent

Exclusion Criteria:

* Pregnancy and/or lactation
* Acute and life-threatening illness (instable angina pectoris, acute pulmonary arterial embolism, myocardial infarction, etc.)
* Any contraindication to undergo thoracoscopy (e.g. anticoagulation therapy which cannot be discontinued for the procedure)
* Any medical, psychological or other condition impairing the patient's ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population for selection of potential study participants is comprised of clinical routine patients presenting with (suspected malignant) pleural effusion. These patients must have an indication for pleural puncture. The cause and nature of the pleural effusion at this time point will be unknown in many cases. To establish this, further diagnostic procedures are required. Only patients with confirmed diagnosis of non-small cell lung cancer will be included in the data analysis.
  A patient in whom suspicion of pleural manifestation of lung cancer is not confirmed, will be considered a screening failure and thus excluded from the study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Winfried J Randerath, Prof. Dr., Principal Investigator — Wissenschaftliches Institut Bethanien e.V
Locations (1):
- Wissenschaftliches Institut Bethanien e. V., Solingen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hagmeyer L, Schafer S, Engels M, Pietzke-Calcagnile A, Treml M, Herkenrath SD, Heldwein M, Hekmat K, Matthes S, Scheel A, Wolf J, Buttner R, Randerath W. High sensitivity of PD-L1 analysis from pleural effusion in nonsmall cell lung cancer. ERJ Open Res. 2021 Mar 22;7(1):00787-2020. doi: 10.1183/23120541.00787-2020. eCollection 2021 Jan. PMID 33778051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical routine patients presenting with (suspected malignant) pleural effusion and indication for pleural puncture were considered for enrollment. Patients with confirmed malignancy of pleural effusion were actually enrolled.
Groups:
- Malignant Pleural Effusion: Patients with confirmed malignant pleural effusion
Period: Overall Study
Arm/Group | Malignant Pleural Effusion
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: patients with confirmed diagnosis of non-small cell lung cancer
Arm/Group | Malignant Pleural Effusion
Number analyzed (Participants) | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72.5 [62.8 to 76.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 50
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 25.7 [23.2 to 28.5]
smoking status [Count of Participants; unit: Participants]
  never | 7
  ex-smoker | 28
  current smoker | 15
Histology Type [Count of Participants; unit: Participants]
  NSCLC - Adeno carcinoma | 33
  NSCLC - Squamous cell carcinoma | 7
  NSCLC - large-cell neuroendocrine carcinoma | 1
  SCLC | 4
  SCLC + Adeno carcinoma | 1
  Non-Hodgkin Lymphoma | 1
  Sarcomatoid Mesothelioma | 1
  Ambiguous histology | 2
Cancer Stage (UICC 8th ed.) [Count of Participants; unit: Participants]
  IA2 | 1
  IB | 1
  IIB | 3
  IIIA | 2
  IIIB | 2
  IVA | 24
  IVB | 15
  Unknown | 1
  III-IV (IMIG classification) | 1

OUTCOME MEASURES:

1. Primary Outcome: PD-L1 Prevalence IHC
Description: Number/prevalence of PD-L1-positive patients according to immunohistochemistry (IHC) of pleural biopsy.
Time Frame: At baseline
Population: Thoracoscopy was performed in all fifty patients. PD-L1 analysis of pleural tissue was indicated in all samples with evidence of tumor cells (n=40), excluding cases with small-cell lung cancer (n=2). Mainly due to insufficient sample material (low tumor cell count) (n=3), PD-L1 analysis could actually be performed in 35 pleural tissue cases.
Measure: Count of Participants; unit: Participants
Groups:
- Number of PD-L1-positive Samples in IHC: For the assessment of potentially therapy-relevant PD-L1 expression levels, two different threshold levels of PD-L1 expression were considered as per the differing approval status (TPS ≥50% and TPS≥1%). Regarding detection of malignancy and PD-L1-positivity, results were defined as negative where the tests were not feasible or in case of inconclusive findings.
Arm/Group | Number of PD-L1-positive Samples in IHC
Number analyzed (Participants) | 35
Participants
  PD-L1 expression with a TPS ≥ 1% was defined as PD-L1-positive: PD-L1 positive | 21
  PD-L1 expression with a TPS ≥ 1% was defined as PD-L1-positive: PD-L1 negative | 14
  PD-L1 expression with a TPS ≥ 50% was defined as PD-L1-positive: PD-L1 positive | 8
  PD-L1 expression with a TPS ≥ 50% was defined as PD-L1-positive: PD-L1 negative | 27

2. Primary Outcome: PD-L1 Prevalence ICC
Description: Number/prevalence of PD-L1-positive patients according to immunocytochemistry (ICC) of pleural aspirate
Time Frame: At baseline
Population: Pleural puncture was performed in all fifty patients. PD-L1 analysis of pleural effusion was indicated in all samples with evidence of tumor cells (n=36), excluding cases with small-cell lung cancer (n=3). Mainly due to insufficient sample material (low tumor cell count) (n=7) or technical issue (n=1), PD-L1 analysis could actually be performed in 25 pleural effusion cases.
Measure: Count of Participants; unit: Participants
Groups:
- Number of PD-L1-positive Samples in ICC: For the assessment of potentially therapy-relevant PD-L1 expression levels, two different threshold levels of PD-L1 expression were considered as per the differing approval status (TPS ≥50% and TPS≥1%). Regarding detection of malignancy and PD-L1-positivity, results were defined as negative where the tests were not feasible or in case of inconclusive findings.
Arm/Group | Number of PD-L1-positive Samples in ICC
Number analyzed (Participants) | 25
Participants
  PD-L1 expression with a TPS ≥ 1% was defined as PD-L1-positive: PD-L1 positive | 19
  PD-L1 expression with a TPS ≥ 1% was defined as PD-L1-positive: PD-L1 negative | 6
  PD-L1 expression with a TPS ≥ 50% was defined as PD-L1-positive: PD-L1 positive | 13
  PD-L1 expression with a TPS ≥ 50% was defined as PD-L1-positive: PD-L1 negative | 12

3. Primary Outcome: PD-L1 Detection in Pleural Effusion Based on All Cases With Successful PD-L1 Analysis
Description: Based on all cases where PD-L1 analysis was indicated and sucessful (i.e. giving definite results), the immunocytochemistry analysis of PE was compared with the immunohistochemistry analysis of pleural tissue.Two different alternatives were calculated:
  * PD-L1 expression with a TPS ≥50% was defined as PD-L1-positive.
  * PD-L1 expression with a TPS ≥1% was defined as PD-L1-positive.
Time Frame: At baseline
Measure: Number (95% Confidence Interval); unit: percent
Groups:
- Sensitivity and Specificity of PD-L1 Detection in Pleural Effusion (TPS ≥50%): Sensitivity and specificity of PD-L1 detection in pleural effusion. PD-L1 expression with a TPS ≥50% was defined as PD-L1-positive.
- Sensitivity and Specificity of PD-L1 Detection in Pleural Effusion (TPS ≥1%): Sensitivity and specificity of PD-L1 detection in pleural effusion. PD-L1 expression with a TPS ≥ 1% was defined as PD-L1 positive.
Arm/Group | Sensitivity and Specificity of PD-L1 Detection in Pleural Effusion (TPS ≥50%) | Sensitivity and Specificity of PD-L1 Detection in Pleural Effusion (TPS ≥1%)
Number analyzed (Participants) | 21 | 21
percent
  Sensitivity | 100 [46 to 100] | 86 [56 to 97]
  Specificity | 63 [36 to 84] | 43 [12 to 80]
  positive predictive value | 45 [18 to 75] | 75 [47 to 92]
  negative predictive value | 100 [66 to 100] | 60 [17 to 93]

4. Secondary Outcome: PD-L1 Detection in Pleural Effusion Based on All Cases With Indication for PD-L1 Analysis
Description: Based on all cases where PD-L1 analysis was indicated, the immunocytochemistry analysis of PE was compared with the immunohistochemistry analysis of pleural tissue.Two different alternatives were calculated:
  * PD-L1 expression with a TPS ≥50% was defined as PD-L1-positive.
  * PD-L1 expression with a TPS ≥1% was defined as PD-L1-positive. In both instances, cases where PD-L1 analysis could not be performed were defined as negative.
Time Frame: At baseline
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Sensitivity and Specificity of PD-L1 Detection in Pleural Effusion (TPS ≥50%) | Sensitivity and Specificity of PD-L1 Detection in Pleural Effusion (TPS ≥1%)
Number analyzed (Participants) | 31 | 31
percent
  Sensitivity | 71 [30 to 95] | 71 [44 to 89]
  Specificity | 71 [49 to 87] | 64 [36 to 86]
  positive predictive value | 42 [16 to 71] | 71 [44 to 89]
  negative predictive value | 89 [65 to 98] | 64 [36 to 86]

5. Secondary Outcome: Tumor Cell Detection in Pleural Effusion
Description: Comparing the immunocytochemistry (ICC) analysis of pleural effusion concerning the detection of malignant tumor cells as compared to the immunohistochemistry analysis of pleural tissue. Seven cases of ICC analysis with inconclusive results were defined as negative.
Time Frame: At baseline
Measure: Number (95% Confidence Interval); unit: percent
Groups:
- Sensitivity and Specificity of Tumor Cell Detection: Sensitivity and specificity of tumor cell detection in pleural effusion. Seven cases of ICC analysis with inconclusive results defined as negative.
Arm/Group | Sensitivity and Specificity of Tumor Cell Detection
Number analyzed (Participants) | 50
percent
  Sensitivity | 83 [67 to 89]
  Specificity | 70 [35 to 92]
  positive predictive value | 92 [76 to 98]
  negative predictive value | 50 [24 to 76]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | NSCLC With Pleural Effusion
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

LIMITATIONS AND CAVEATS:
The fact that the PE did not always yield enough material for a comprehensive immunocytochemistry evaluation including PD-L1 analysis, constitutes an important limitation, in part leading to inconclusive results regarding malignancy. This may be due to a low rate of cells scaling off from the pleural lesion and/or a low rate of migration of tumor cells into the pleural fluid.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT02855281/Prot_SAP_000.pdf